CLINICAL TRIAL: NCT03474523
Title: Effectiveness of Diathermy-Radiofrecuency Compared With Cavitation in Cellulitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Ines Carmona Barrientos, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fisioterapia Bahía
Record Dates: First submitted 2018-02-08; First posted 2018-03-22 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cellulitis
Keywords: radio frequency diathermy; cavitation; ultrasound; edemato-fibrosclerotic panniculopathy; cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled longitudinal experimental study
Who Masked: Participant, Outcomes Assessor
Masking Description: external evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental or Diathermy-Radiofrecuency (Experimental): All patients are given a Combined Physiotherapy Protocol (CPP) consisting of: Diathermy-Radiofrecuency (manual 70% intensity of about 40-43º resistive modality for about 30 minutes and authomatic capacitive modality for about 10 minutes) and application of Presotherapy (intensity 35%, compression 35seg, pause 15 seg, speed 9, for about 30 minutes). Non-invasive treatment
  Interventions: Other: Experimental group
- Control or Cavitation (Active Comparator): All patients are given a Combined Physiotherapy Protocol (CPP) consisting of: Cavitation (plane electrode for about 30 minutes and focal electrode for about 10 minutes) at 70% intensity and application of Presotherapy (intensity 35%, compression 35seg, pause 15 seg, speed 9, for about 30 minutes). Non-invasive treatment
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Cavitation: 70% intensity, 30 minutes apply plane electrode and 10 minutes focal electrode.
  Presotherapy: 30 minutes application of 35% intensity, compression 35seg, pause 15seg, speed 9
  Arms: Experimental or Diathermy-Radiofrecuency
Other: Control group — Diathermy-Radiofrecuency: 30 minutes at 70% intensity (40-43ºC) in manual resistive modality and 10 minutes in automatic capacitive modality.
  Presotherapy: 30 minutes application of 35% intensity, compression 35seg, pause 15seg, speed 9
  Arms: Control or Cavitation

SUMMARY:
The aim of the present study is to value the effectiveness of Diathermy-Radiofrecuency treatment compared to Cavitation treatment in woman with cellulitis.

DETAILED DESCRIPTION:
The edemato-fibrosclerotic panniculopathy is a segmental disease and lipodystrophy, this disease is localized in subcutaneous connective tissue which is influenced by venous and lymphatic system, when these systems are affected. The secondary vasomotor dysfunction to failure sympathetic nervous system influence on this disease too.

Usually it affects women, influencing their physical and psychological well-being.

The Aesthetic Physiotherapy, known as Aesthetics Plastic and Restorative Physiotherapy, is in their beginnings, there are little studies which present this pathology from the physiotherapy perspective. The investigators believe that their research could make some progress in this matter.

The search found very few clinical trials of scientific rigor about radio frequency and cavitation, and The investigators didn't find studies that compare both. Both treatments show effectiveness in improving the appearance of cellulite, so it would be a good idea compare them and see the most effective.

The investigators are trying to compare the effectiveness of both techniques and the investigators consider innovative and with added value to investigate something that we haven´t found in the reviewed literature.

The investigators choose 20 women randomly, 40 sample subjects, between 18-40 years old. These women must keep the inclusion criteria.

The participants attend a first date where the investigators collect the necessary data, and they are valued before and after the treatment (perimetry, photographic, Nürnberger and Müller scale, weight, height, BMI).

Then each patient receive treatment, seven non-consecutive sessions Diathermy-Radiofrequency on one leg (gluteal zone, internal and lateral zone, posterior and anterior zone) and other 7 sessions of Cavitation in the other leg, and Presotherapy in both legs.

The investigators also advice the participants about their diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female
* UCA comunity
* Age 18-40 years
* Cellulite grade I, II, III (Nürnberg&Müller clasification)
* Compliance of study timing
* Acceptance of informed consent and signature of study authorization

Exclusion Criteria:

* Pacemaker, heart diseases, epilepsy,
* pregnancy, lactation, last year postpartum, menstrual cycle alterations, climacteric, perimenopause
* chronic disease, hormonal or circulatory disorder, neoplasia process
* inflammation, infection, active acne, open wound in the treatment area
* BMI above 27 Kg/m2, obesity, lipoedema, oedema, circulatory problems
* Metal implants, prosthesis, intrauterine devices
* Evolutive diseases
* Severe Artheryal hipertension
* High cholesterol levels or non-controlled triglycerides
* Weight fluctuation above 2 kg in the last six months
* Drinking more than two daily alcoholic drinks
* Pharmacological treatment during study: anti-inflammatory, esthetical, cosmetical or dietetic treatment
* Previous treatment of the studies areas in the last year
* Surgery intervention in studies areas

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — PEFE has a greater incidence within women
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Decrease in perimeter measures | At the begining and at the end of the treatment after seven weeks
  measuring tape

SECONDARY OUTCOMES:
Changes in body mass index | At the begining and at the end of the treatment after seven weeks
  Calculation of the body mass index
Changes in weight | At the begining and at the end of the treatment after seven weeks
  Weighing machine
Physical activity evaluation | At the begining and at the end of the treatment after seven weeks
  IPAQ questionnaire
Degree of cellulitis | At the begining and at the end of the treatment after seven weeks. This scale measures the level of cellulite and takes the values of 0-3, being 0 the value where there is no cellulite and 3 the most serious stage of cellulite.
  Nürberger and Müller's scale

CONTACTS AND LOCATIONS:
Overall Officials: Carmona I. Barrientos, Dra, Principal Investigator — University of Cadiz
Locations (1):
- Faculty of Nursing and Physiotherapy. University of Cadiz, Cadiz, Spain